CLINICAL TRIAL: NCT01456728
Title: Efficacy of Dietary Supplementation With Lactobacillus Reuteri ProGastria in Helicobacter Pylori-infected Adult Subjects Treated Only With Proton Pump Inhibitors
Brief Title: Lactobacillus Reuteri ProGastria in Helicobacter Pylori-infected Adult Subjects on Proton Pump Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St Marina University Hospital, Varna, Bulgaria (Other)
Responsible Party: Principal Investigator, Iskren Kotzev, Professor Iskren Kotzev MD, PhD, MSc, St Marina University Hospital, Varna, Bulgaria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34/30.06.2011
Record Dates: First submitted 2011-10-07; First posted 2011-10-21 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Progastria; Lactobacillus reuteri; omeprazole; triple therapy; probiotic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Progastria (Experimental): One chewable tablet of the study product is to be taken once per day giving a dose of L. reuteri of 2x108 CFU/day together with omeprazole 2x20mg. The study product and omeprazole will be taken daily for 28 consecutive days.
  Interventions: Dietary Supplement: Progastria
- Placebo (Placebo Comparator): The placebo will have identical appearance and taste with the study product only lacking the bacteria. All subjects from this group will receive 2 x 20 mg omeprazole per day and Placebo 1 chewable tablet per day for 28 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Progastria — All subjects will receive 2 x 20 mg omeprazole per day for 28 days.
  L. reuteri ProGastria will be delivered at a dose of 1x108 CFU of 2 strains of L. reuteri giving a final dose of L. reuteri of 2x108 CFU. One chewable tablet is to be taken once per day giving a dose of L. reuteri of 2x108 CFU/day. This dose of L. reuteri has been shown to be effective in a series of conditions earlier, including inhibition of H. pylori in humans, and is considered the optimal dose. The study products will be taken daily for 28 consecutive days.
  Arms: Progastria
Dietary Supplement: Placebo — The placebo will have identical in appearance and taste with the active study product only lacking the bacteria. It will be prescribed the same way as ProGastria: omeprazole 2x20mg and Placebo 1 tablet per day for 28 consecutive days
  Arms: Placebo

SUMMARY:
The purpose of the study is to confirm that simultaneous use of L. reuteri ProGastria and omeprazole for 28 days can eradicate H. pylori in humans in the absence of antibiotics.

DETAILED DESCRIPTION:
Helicobacter pylori colonises an estimated 50% of the world´s population. Despite clear clinical guidelines on the treatment of this infection there is a drive to find alternative ways to control this infection in a wider perspective without the complications of induction of antibiotic resistance in the pathogen. A good alternative is to use probiotics.

Lactic acid bacteria and in particular lactobacilli have been studied for their effects in humans infected with H. pylori with some success in reducing the infection load. Studies using supplementation with L. reuteri in both symptomatic and non-symptomatic H. pylori-infected subjects show a clear reduction of infection load after 4 weeks of use and this was concomitant with a reduction in symptoms associated with the infection. Further, dietary supplementation with L. reuteri during and after the period of H. pylori eradication therapy has also been shown to reduce the side effects of this therapy without affecting the degree of eradication.

ELIGIBILITY:
Inclusion Criteria:

* Infection with H. pylori defined using the 13C-urea breath test
* Non-ulcer dyspepsia
* No earlier eradication therapy for H. pylori infection
* Written informed consent
* Stated availability throughout the entire study period
* Mental ability to understand and willingness to fulfil all the details of the protocol.

Exclusion Criteria:

* Duodenal or gastric ulcer
* MALT lymphoma
* Gastric resection (at any time)
* First level relatives of gastric cancer patients
* Absence of GI symptoms
* Use of NSAIDs, aspirin or other anti-inflammatory drugs within 1 week (for occasional use) or 3 weeks (for chronic use) of inclusion
* Use of oral antibiotics and/or PPIs and/or H2-antagonists during the 2 weeks prior to ingestion of the study product
* Pregnancy
* Participation in other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Increased number of H. pylori positive subjects treated with L. reuteri-ProGastria for 28 days who are negative for H. pylori after the treatment compared to placebo | 1 year
  Increase in the number of subjects with treatment success after 28 days of treatment with omeprazole + L. reuteri ProGastria compared to those given omeprazole + placebo will prove treatment success defined as the absence of H. pylori infection on Day 29. This is measured as a significant reduction in gastrointestinal symptoms (according to a validated GSRS score) and a negative stool antigen test for H. pylori infection.

SECONDARY OUTCOMES:
Increased number of subjects from the ProGastria group compared to the placebo group with a maintained absence of H.pylori infection up to 2 months after completed treatment | 1 year
  This outcome measure will be proven when there is evidence of fewer patients in the L. reuteri ProGastria treatment success group with demonstrated presence of H. pylori infection, measured as UBT on Day 90 compared to the placebo treatment success group.
Number of patients with amelioration of gastrointestinal symptoms in H. pylori-infected subjects treated with ProGastria compared to placebo. | 1 year
  This is achieved by following reduced gastrointestinal symptom scores using GSRS validated scoring system at days 14, 28 and 90 in L. reuteri ProGastria treated subjects compared to placebo.
Confirmation that L. reuteri +omeprazole could improve eradication rates of H. pylori using triple therapy | 1 year
  This measure will be done by assesing the absence of H. pylori infection on Day 90 measured as a negative outcome in UBT in the L. reuteri ProGastria treatment failure group compared to the placebo treatment failure group

CONTACTS AND LOCATIONS:
Overall Officials: Iskren Kotzev, MSc, Principal Investigator — Head, Clinik of Gastroenterology
Locations (1):
- Department of Gastroenterology and Hepatology, St Marina University Hospital, Varna, Bulgaria, Bulgaria